CLINICAL TRIAL: NCT04772924
Title: Is Prolonged Fasting Safe in Patients Who Underwent Percutaneous Coronary Intervention More Than One Year Earlier?
Brief Title: Long-term Fasting in Patients With a History of PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IR.SUMS.MED.REC.1398.465
Record Dates: First submitted 2021-02-19; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
Keywords: prolonged fasting; percutaneous coronary angioplasty; major adverse cardiac events
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fasting group (Experimental): those preferred to take long time fasting
  Interventions: Behavioral: fasting
- non fasting (Active Comparator): those preferred not to take fasting
  Interventions: Behavioral: not fasting

INTERVENTIONS:
Behavioral: fasting — more than 12 hour of fasting as ceremony of Ramadan
  Arms: fasting group
Behavioral: not fasting — preferred not to take long term fasting
  Arms: non fasting

SUMMARY:
Patients in this prospective cohort study were selected if they had a history of PCI more than 1 year previously. 405 patients were divided based on their preferences to fasting and non fasting and after 1 month of fasting major adverse cardiovascular events were measured

DETAILED DESCRIPTION:
Between 18 March 2019 and 18 April 2020, patients seen at Professor Kojuri Cardiovascular Clinic in Shiraz, Iran (email:kojurij@yahoo.com, webpage: http://kojuriclinic.com) for their annual check-up were selected. We explained the research project to them, and volunteers were selected. Patients were assigned to the fasting or non-fasting group according to their preference. All volunteers were informed about the details of this research, and provided their written informed consent. Patients who declined to participate in the study were excluded.

Patients were instructed how to divide their medication across the two daily meals before dawn and after sunset during the month of Ramadan. We informed patients to immediately stop fasting and consult the clinic if they experienced any signs of cardiovascular disease, including shortness of breath, chest pain, or palpitations. At the end of Ramadan, patients were contacted by telephone and asked about their symptoms, including chest pain and dyspnea, hospitalization, and MACE. The MACE were defined as acute myocardial infarction, hospitalization due to congestive heart failure, new-onset atrial fibrillation, stroke, or cardiac arrest [19, 20]. Symptomatic patients were referred to the clinic for cardiovascular examination.

The study was double-blinded. To blind the researchers, the clinic secretary contacted the patients and asked them not to specify their group (fasting or non-fasting), and then passed the phone to the researcher. We used alphabetical order in each group to blind the statisticians. Patients who fasted during Ramadan were designated with the letter X, and patients who did not fast during Ramadan were designated with the letter Y.

For statistical analyses we used IBM SPSS software version 25. We used the chi-squared test to compare categorical variables and Student's t-test to compare the mean values of continuous variables. The Mann-Whitney U test and Kruskal-Wallis test were used for nonparametric variables.

ELIGIBILITY:
Inclusion Criteria:

* history of PCI, and a minimum of 1 year between angioplasty and enrollment in this study

Exclusion Criteria:

* Heart failure (ejection fraction <50 %)
* Advanced kidney failure (glomerular filtration rate <60 mL/min
* Unsuccessful revascularization
* Coronary artery bypass graft
* Liver cirrhosis
* Any acute conditions such as infection
* Needed repetitive treatment
* Diabetes who were on insulin treatment

Ages: 53 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The number of participant with major adverse cardiovascular event | 1 month

SECONDARY OUTCOMES:
Dyspnea | 1 month
  Grade of dyspnea was measured based on patient report, based on New York heart association class, 1 no dyspnea, 2 dyspnea at heavy exertion, 3 dyspnea at sub maximal exertion, 4 dyspnea at rest
Angina based on patient report, based on Canadian heart class | 1 month
  1 no chest pain, 2 chest pain at maximal exercise, 3 chest pain at submaximal exercise, 4 chest pain at rest

CONTACTS AND LOCATIONS:
Locations (1):
- Professor kojuri cardiology clinic, Shiraz, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: No